CLINICAL TRIAL: NCT03084978
Title: Randomized Prospective Study in Transcatheter Aortic Valve Replacement Patients- Conscious Sedation VS. General Anesthesia Examining the Effect on Operative Time
Brief Title: Conscious Sedation vs General Anesthesia in TAVR Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never approved by the IRB
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-7021
Record Dates: First submitted 2017-01-25; First posted 2017-03-21 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Anesthesia, General; Conscious Sedation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (Active Comparator): Subjects will undergo general anesthesia with endotracheal intubation.
  Interventions: Procedure: General Anesthesia
- Conscious Sedation (Experimental): Subjects will undergo conscious sedation anesthesia.
  Interventions: Procedure: Conscious Sedation

INTERVENTIONS:
Procedure: General Anesthesia — General anesthesia by standard endotracheal intubation.
  Arms: General Anesthesia
Procedure: Conscious Sedation — Conscious sedation
  Arms: Conscious Sedation

SUMMARY:
This is a randomized controlled trial investigating the effect of general anesthesia versus conscious sedation on operative times in patients undergoing transcatheter aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, signed Health Insurance Portability and Accountability Act (HIPAA) documentation)
2. Age over 18 years of age.
3. Women of child bearing age must have a negative urine or serum pregnancy test.
4. Clinical indication for a transfemoral aortic valve replacement.
5. English or Spanish speaking
6. No evidence of neurological impairment as defined by a NIHSS ≤ 1 and modified Rankin scale (mRS) ≤ 2 within 7 days prior to randomization.

Exclusion Criteria:

1. BMI > 40
2. Diagnosis of severe obstructive sleep apnea based on previous polysomnography, with severe defined as an apnea-hypopnea index (AHI) >30 episodes/hr.
3. High risk for aspiration such as severe esophageal disease (e.g. achalasia, gastroparesis, etc).
4. Inability to lie supine for more than 30 minutes.
5. Marginal femoral vessels with concern for possible conversion to transapical or transaortic access.
6. Patient refusal
7. Patient involved in another research study
8. Psychiatric condition precluding ability to provide informed consent
9. History of clinical stroke within 3 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Time-on-table | <1 day
  * time to patient on table to surgical drapes down
  * time to patient on table to when deemed safe for transport by anesthesiologist and surgeon

SECONDARY OUTCOMES:
Number of patients with serious adverse events | within 30 days
  * deaths
  * conversion from sedation to intubation
  * hypersensitivity reactions
Length of stay | within 30 days
  * ICU length of stay (days)
  * Hospital length of stay (days)
Readmissions | within 30 days
  Number of patients readmitted within 30 days of initial procedure
Number of Patients with Valve Complications | within 30 days
  * paravalvular leak on echocardiogram
  * pacemaker requirement
  * vascular complications requiring reintervention
  * post-procedure requiring valve dilation
Contrast usage | <1 day
  Amount of contrast used in mL for procedure
Fluoroscopy time | <1 day
  Amount of time fluoroscopy used

OTHER OUTCOMES:
Post-procedure Complications | within 30 days
  * TIA or Stroke
  * Myocardial Infarction
  * Bleeding
  * Infection
Quality of Life | Procedure start to 30 days
  Kansas City Cardiomyopathy Questionnaire at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph DeRose, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brecker SJ, Bleiziffer S, Bosmans J, Gerckens U, Tamburino C, Wenaweser P, Linke A; ADVANCE Study Investigators. Impact of Anesthesia Type on Outcomes of Transcatheter Aortic Valve Implantation (from the Multicenter ADVANCE Study). Am J Cardiol. 2016 Apr 15;117(8):1332-8. doi: 10.1016/j.amjcard.2016.01.027. Epub 2016 Jan 28. PMID 26892451